CLINICAL TRIAL: NCT06531772
Title: Characteristics and Outcomes of TB and HIV Co-infections
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Assistant Professor of Chest Diseases, Assiut University
Other Study IDs: WG72024
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Human Immunodeficiency Virus; Mycobacterium Tuberculosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Antitubercular Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tuberculosis without HIV
  Interventions: Drug: Antitubercular Agents
- Tuberculosis with HIV Coinfection
  Interventions: Drug: Antitubercular Agents

INTERVENTIONS:
Drug: Antitubercular Agents — Full regimen of antitubercular drugs for 6 month period or longer as justified by patient condition

SUMMARY:
People Living with HIV (PLHIV) are prone to several opportunistic infections depending on the degree of immunosuppression as well as infections prevalent in their geographic area/country. These include a wide variety of mycobacterial diseases, fungal infections, bacterial pneumonias, pneumocystis jirovecii pneumonia, cryptococcal infections, toxoplasmosis etc.

Tuberculosis remains the most common opportunistic infection in the developing countries like South Africa and India.

HIV and tuberculosis (TB) are two of the most challenging infections faced by the humanity. HIV is the most important risk factor for progression of latent Mycobacterium tuberculosis (MTB) to active disease. The most common cause of death among PLHIV is tuberculosis. These two infections place immense burden on health care systems worldwide. During the last two decades, sustained research and public health initiatives on prevention and therapeutic advances have allayed morbidity and mortality due to HIV and TB to a large extent, however more needs to be done.

Globally, an estimated 10 million people fell ill with TB and an estimated 1.4 million people died of TB in 2018 (1.2 million among HIV negative and 251 000 among HIV positive people). There were around 37.9 million PLHIV worldwide in 2018.

In the pre-antiretroviral therapy (ART) era, nearly one-third of HIV/AIDS (acquired immune deficiency syndrome) related deaths were due to TB. Wider availability of ART has reduced the mortality of HIV-associated TB significantly, but it still remains high compared to HIV-uninfected individuals. The mortality risk with HIV TB coinfection accounts for approximately 25% of global HIV/AIDS deaths every year.

This study aims to investigate characteristics and outcomes of TB and HIV co-infections in Upper Egypt.

DETAILED DESCRIPTION:
People Living with HIV (PLHIV) are prone to several opportunistic infections depending on the degree of immunosuppression as well as infections prevalent in their geographic area/country. These include a wide variety of mycobacterial diseases, fungal infections, bacterial pneumonias, pneumocystis jirovecii pneumonia, cryptococcal infections, toxoplasmosis etc.

Tuberculosis remains the most common opportunistic infection in the developing countries like South Africa and India.

HIV and tuberculosis (TB) are two of the most challenging infections faced by the humanity. HIV is the most important risk factor for progression of latent Mycobacterium tuberculosis (MTB) to active disease. The most common cause of death among PLHIV is tuberculosis. These two infections place immense burden on health care systems worldwide. During the last two decades, sustained research and public health initiatives on prevention and therapeutic advances have allayed morbidity and mortality due to HIV and TB to a large extent, however more needs to be done.

Globally, an estimated 10 million people fell ill with TB and an estimated 1.4 million people died of TB in 2018 (1.2 million among HIV negative and 251 000 among HIV positive people). There were around 37.9 million PLHIV worldwide in 2018.

In the pre-antiretroviral therapy (ART) era, nearly one-third of HIV/AIDS (acquired immune deficiency syndrome) related deaths were due to TB. Wider availability of ART has reduced the mortality of HIV-associated TB significantly, but it still remains high compared to HIV-uninfected individuals. The mortality risk with HIV TB coinfection accounts for approximately 25% of global HIV/AIDS deaths every year.

This study aims to investigate characteristics and outcomes of TB and HIV co-infections in Upper Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory diagnosis of TB-HIV co-infection

Exclusion Criteria:

* Patients refusing to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients visiting Tuberculosis clinic - Assiut university hospitals for receiving antitubercular medicines will be divided into 2 groups either; A- Tuberculosis Cases, or B- Tuberculosis-HIV coinfection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate for tuberculosis infection | 6 months
  complete cure from tuberculosis infection assessed by sputum conversion, general condition improvement and radiological improvement.

SECONDARY OUTCOMES:
pulmonary complications associated with tuberculosis in both groups | 1 year
  Superimposed pneumonia, opportunistic infection, pneumothorax, respiratory failure

CONTACTS AND LOCATIONS:
Overall Officials: Waleed MD Gamal Elddin Khaleel, Ass. Prof., Principal Investigator — Assiut University
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khadka P, Thapaliya J, Basnet RB, Ghimire GR, Amatya J, Rijal BP. Diagnosis of tuberculosis from smear-negative presumptive TB cases using Xpert MTB/Rif assay: a cross-sectional study from Nepal. BMC Infect Dis. 2019 Dec 30;19(1):1090. doi: 10.1186/s12879-019-4728-2. PMID 31888522
- [Background] Agarwal U, Kumar A, Behera D. Profile of HIV associated tuberculosis at a tertiary institute in setting of free anti-retroviral therapy. J Assoc Physicians India. 2009 Oct;57:685-90. PMID 20329424
- [Background] Yang Q, Han J, Shen J, Peng X, Zhou L, Yin X. Diagnosis and treatment of tuberculosis in adults with HIV. Medicine (Baltimore). 2022 Sep 2;101(35):e30405. doi: 10.1097/MD.0000000000030405. PMID 36107594